CLINICAL TRIAL: NCT04247945
Title: Co-transplantation of Mesenchymal Stromal Cells in Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Co-transplantation of MSC in the Setting of Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Professor of Hematology, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSC-SCT-03
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSC (No Intervention)
- MSC+HSC (Experimental)
  Interventions: Biological: Cotransplant with MSCs

INTERVENTIONS:
Biological: Cotransplant with MSCs — Co-transplantation of MSCs during allogeneic HSCT
  Arms: MSC+HSC

SUMMARY:
Mesenchymal stem cells (MSCs) are known to exhibit immunomodulatory, anti-inflammatory, and pro-angiogenic properties, and therefore have the potential to improve the outcome of allogeneic hematopoietic stem cell transplantation (allo-HSCT) .The study is aimed to identify and evaluate the potential benefits of MSCs infusion during allogeneic HSCT, with regard to the engraftment, graft versus host disease (GVHD), post-transplant relapse and survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged <65 years
* Willing to transplant
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of MSCs.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | up to 2 years after HSCT

SECONDARY OUTCOMES:
Cumulative Incidence of Graft-versus Host Disease | up to 2 years after HSCT
Incidence of Systemic Infections | up to 2 years after HSCT
Mean Time to Engraftment | Baseline to engraftment, assessed minimally 28 days post transplant
Transplant-Related Mortality | up to 1 months after HSCT
Rates of Relapse | up to 2 years after HSCT

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital,Fujian Medical University, Fuzhou, Fujian, China